CLINICAL TRIAL: NCT02073760
Title: Optimizing Prevention of Healthcare-Acquired Infections After Cardiac Surgery (HAI)_2
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Dr. Donald Likosky, Associate Professor, University of Michigan
Other Study IDs: HAI_Umich_2; 2004-0428 (Other: UMichigan's IRB)
Record Dates: First submitted 2014-02-21; First posted 2014-02-27 (Estimated); Last update posted 2018-10-22 (Actual); Status verified 2018-10

CONDITIONS: Cardiovascular Disease; Healthcare Associated Infectious Disease; Sternal Superficial Wound Infection; Deep Sternal Infection; Mediastinitis; Thoracotomy; Conduit Harvest or Cannulation Site; Sepsis; Pneumonia
Keywords: Healthcare acquired infections; Cardiac Surgery; Sternal Superficial Wound Infection; Deep Sternal Infection; Mediastinitis; Thoracotomy; Conduit harvest or cannulation site; Sepsis; Pneumonia
MeSH Terms: conditions — Cardiovascular Diseases; Cross Infection; Mediastinitis; Sepsis; Pneumonia | interventions — Caregivers

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Infection Prevention Experts: Adult caregivers of cardiac surgery patients (e.g. surgeons, nurses, infection preventionists) and administrators
  Interventions: Other: There is no intervention. The investigators are interviewing cardiac surgery staff with knowledge of infection prevention.

INTERVENTIONS:
Other: There is no intervention. The investigators are interviewing cardiac surgery staff with knowledge of infection prevention. — The investigators will conduct tape recorded interviews with hospital staff about infection prevention.
  Other Names: Caregivers

SUMMARY:
The investigators will conduct qualitative interviews of hospital personnel regarding HAI prevention practices, and use coded data from these interviews to assist in developing standardized practices.

DETAILED DESCRIPTION:
More than 400,000 coronary artery bypass grafting (CABG) procedures are performed every year in the United States (U.S.). Patients undergoing CABG surgery are at risk for a number of adverse sequelae, many of which impact survival and contribute to overall health-care costs. Healthcare-acquired infections (HAIs), including pneumonia and superficial and deep sternal wound infections, occur among 16% of CABG patients and elevate a patient's risk of mortality and add excess upfront and long-term expenditures to the health care system.

A number of barriers prevent wide-scale improvements in HAl rates within the setting of CABG surgery. While a number of HAl prophylaxis measures have been developed, these measures do not fully encompass the set of practices that may impact a patient's risk of HAl. Identifying cardiac surgery specific risk factors would serve as the foundation for targeted quality improvement strategies. In the absence of definitive data concerning best practices, HAl prophylaxis is variable across surgeons and institutions, resulting in unnecessary morbidity and cost. Prior work has shown the value of implementing evidence-based protocols in the general intensive care unit setting. To what extent the implementation of cardiac surgery specific standardized practices results in lower HAl rates is uncertain. An understanding of the effectiveness of this approach would certainly assist surgeons and institutions in providing safer care to their patient populations.

Rates of HAIs vary from 0-26% across the 33 institutions performing CABG surgery in Michigan. This application seeks to reduce this rate by identifying and subsequently implementing standardized practices, and evaluating their impact on HAl rates. This study will be based on the prospective data and regional quality improvement activities and infrastructure of the Michigan Society of Thoracic and Cardiovascular Surgeons Quality Collaborative (MSTCVS-QC). The investigators will evaluate the effectiveness of these standardized practices in reducing HAIs regionally and relative to national rates during the same time period.

The investigators will conduct qualitative interviews of hospital personnel regarding HAI prevention practices, and use coded data from these interviews to assist in developing standardized practices.

ELIGIBILITY:
Inclusion Criteria:

* Clinical providers or
* Administrators
* Must work at any of 33 institutions performing cardiac surgery in the state of Michigan

Exclusion Criteria: Under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Clinical providers and administrators working at any of 33 institutions performing cardiac surgery in the state of Michigan
Sampling Method: Non-Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2014-06; Primary Completion 2018-09-29 (Actual); Study Completion 2018-09-29 (Actual)

PRIMARY OUTCOMES:
Preventive Strategies | During the time of the interview
  Preventive strategies currently being conducted at their institution to prevent healthcare-acquired infections.

CONTACTS AND LOCATIONS:
Overall Officials: Donald S Likosky, Ph.D., Principal Investigator — University of Michigan
Locations (1):
- Mstcvs-Qc, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
Only upon invitation and in accordance with our contractual obligations

REFERENCES:
- [Background] Likosky DS, Paone G, Zhang M, Rogers MA, Harrington SD, Theurer PF, DeLucia A 3rd, Fishstrom A, Camaj A, Prager RL; Michigan Society of Thoracic and Cardiovascular Surgeons Quality Collaborative. Red Blood Cell Transfusions Impact Pneumonia Rates After Coronary Artery Bypass Grafting. Ann Thorac Surg. 2015 Sep;100(3):794-800; discussion 801. doi: 10.1016/j.athoracsur.2015.03.089. Epub 2015 Jul 21. PMID 26209489